CLINICAL TRIAL: NCT03385772
Title: The Sphenopalatine Ganglion Block as a Treatment Modality for Post-dural Puncture Headache in the Post-partum Patient
Brief Title: The Sphenopalatine Ganglion Block for Post-dural Puncture Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Mihaela Podovei, Instructor, Harvard Medical School, Staff Anesthesiologist, Department of Anesthesia, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017P002523
Record Dates: First submitted 2017-12-21; First posted 2017-12-28 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Post-Dural Puncture Headache
Keywords: sphenopalatine block
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Sphenopalatine Ganglion Block

STUDY DESIGN:
Intervention Model Description: This is a prospective interventional pilot study of the efficacy of the sphenopalatine ganglion block for treatment of post-dural puncture headache in post-partum women.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Sphenopalatine ganglion block — The patient will be placed supine, with head in sniffing position. Two long cotton-tipped applicators will be soaked in 4% lidocaine for 30 seconds. An anesthesia provider, after visually inspecting each nostril for any sign of deformity or blockage, will perform the block. A cotton tipped applicator will be inserted into one nostril at an angle perpendicular to the face, and will be advanced to the back of the nasopharynx until resistance is met. The procedure will be repeated in the other nostril. If the patient experiences any pain or discomfort, the physician will stop and redirect the applicator. The applicators will be left in place for 10 minutes, and then removed by the anesthesia provider.

SUMMARY:
This study aims to determine the efficacy of the sphenopalatine ganglion block in the treatment of post-dural puncture headache in post-partum women at the Brigham and Women's Hospital by measuring VAS scores at times between 0 and 24 hours after the block. We hypothesize that there will be at least a 50% reduction in VAS scores at 4 hours after performing the sphenopalatine block as compared to baseline VAS scores.

DETAILED DESCRIPTION:
Post-dural puncture headache (PDPH) is a major cause of morbidity in postpartum patients who received neuraxial anesthesia for labor analgesia or cesarean delivery. The headache in PDPH is thought to be due to loss of cerebrospinal fluid causing downward traction on the meninges with parasympathetic ally mediated reflex vasodilation of the meningeal vessels. The epidural blood patch is currently the gold-standard treatment for postdural puncture headache, however it is an invasive procedure with possible risks and complications including bleeding, infection, pain, hematoma, neurologic complications, and repeat dural puncture. Patients are often offered conservative treatment including medications, bed rest, abdominal binders, and fluids for at least 24 hours prior to being offered an epidural blood patch. Once the decision is made to proceed with a blood patch, it may take several hours before the procedure is performed due to staffing issues. We propose that the sphenopalatine ganglion block, a relatively noninvasive procedure which has been used by neurologists as a treatment for a variety of types of headaches, may play a role in the treatment of postdural puncture headache in the obstetric population.The sphenopalatine ganglion is a parasympathetic ganglion located in the pterygopalatine fossa which can be accessed topically through the nose. The proposed mechanism of the sphenopalatine ganglion block is parasympathetic blockade preventing the profound vasodilation associated with the headache after a dural puncture, thus providing the patient with symptomatic relief. While the sphenopalatine ganglion block has been used by neurologists for the treatment of migraines and cluster headaches for years, little is known about its effectiveness in the treatment of post-dural puncture headache in post-partum women. A small case series by Kent et al demonstrated that offering the sphenopalatine ganglion block as a first-line treatment for post-dural puncture headache provided symptomatic relief and reduced the need for epidural blood patch. If the sphenopalatine ganglion block is found to be an effective treatment for post-dural puncture headache in the obstetric population, the block could be offered to patients as a firstline treatment as a way to improve VAS scores, reduce the need for medications with potential side effects, and possibly reduce the need for epidural blood patch.The primary outcome will be change in VAS scores at 4 hours after the sphenopalatine ganglion block. Secondary outcomes will include time to first Fioricet dose after the sphenopalatine ganglion block, presence of nausea at 4 hours, presence of neck pain at 4 hours, presence of visual changes at 4 hours, change in VAS scores at 12 hours, change in VAS scores at 24 hours, and need for epidural blood patch.

ELIGIBILITY:
Inclusion Criteria:

* All postpartum women aged 18-50 who received neuraxial anesthesia for labor or cesarean delivery and are diagnosed with a post-dural puncture headache within 72 hours post-partum will be eligible to participate.

Exclusion Criteria:

* Patients with a history of migraines, chronic headaches, chronic narcotic use, chronic neurological disorder, bleeding disorder, deformity of nasal septum, allergy to local anesthetics, nasal polyps, frequent nosebleeds, those with a diagnosis of pregnancy induced hypertension or pre-eclampsia in the most recent pregnancy, and those with nasal or sinus surgery within the past year will be ineligible to participate.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study is on postpartum women with post dural puncture headache after neuraxial anesthesia for delivery.
Enrollment: 20 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Change in VAS scores for headache at 4 hours after the sphenopalatine ganglion block. | 4 h post-intervention
  measured VAS for headache

SECONDARY OUTCOMES:
Time to first request of medication for symptom control after the sphenopalatine ganglion block, | 24 h
Need for blood patch | 24 h
  performance of epidural blood patch for treatment of PDPH
Presence of nausea, neck pain, visual changes post-intervention | periodic questioning over 24h
  yes/no questions
Symptomatic relief of headache after the block | 24 h
  VAS scores at different time points via pain diaries

IPD SHARING:
Plan to Share IPD: No
All data obtained during this study, both clinical and other data including pain diaries, will be kept confidential. Participants will be de-identified using codes so that the names of the study participants will be known only to the study investigators. No information about the identity of individual subjects will be used for publication. The pain diaries and consent forms will be kept in a locked file cabinet. All study data will be kept on a password-protected computer and only the research investigators will have access to the database.

REFERENCES:
- [Background] Kent S, Mehaffey G. Transnasal sphenopalatine ganglion block for the treatment of postdural puncture headache in obstetric patients. J Clin Anesth. 2016 Nov;34:194-6. doi: 10.1016/j.jclinane.2016.04.009. Epub 2016 May 11. PMID 27687372
- [Background] Nair AS, Rayani BK. Sphenopalatine ganglion block for relieving postdural puncture headache: technique and mechanism of action of block with a narrative review of efficacy. Korean J Pain. 2017 Apr;30(2):93-97. doi: 10.3344/kjp.2017.30.2.93. Epub 2017 Mar 31. PMID 28416992